CLINICAL TRIAL: NCT02678676
Title: An Observational Study of Patient Cohorts Who Previously Received Long-term Treatment With Pioglitazone or Placebo in Addition to Existing Antidiabetic Medications.
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: AD-4833/EC445
Record Dates: First submitted 2016-02-07; First posted 2016-02-10 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pioglitazone: Participants who previously received pioglitazone in the PROactive study (NCT00174993).
  Interventions: Other: No Intervention
- Placebo: Participants who previously received Pioglitazone-matching placebo in the PROactive study (NCT00174993).
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants who previously received Pioglitazone in the PROactive study (NCT00174993).
  Groups: Pioglitazone
Other: No Intervention — Participants who previously received pioglitazone-matching placebo in the PROactive study (NCT00174993).
  Groups: Placebo

SUMMARY:
The purpose of this study was to investigate the mortality and macrovascular morbidity as well as the incidence of malignancies over time, in high-risk diabetic participants who previously received long-term treatment with either pioglitazone or placebo in combination with their usual medication for glycaemic management.

DETAILED DESCRIPTION:
This was a European,multicenter,observational study of participants who were previously treated with pioglitazone or placebo in addition to their existing anti diabetic medication. This 10-year observational study was conducted as a follow-up of PROactive study (NCT00174993) to investigate the CV and macrovascular effects observed with pioglitazone over time during PROactive.In this study,high risk T2DM patients previously enrolled in PROactive were analyzed for long-term incidence,nature, and pattern of all malignancies in pioglitazone and placebo-treated groups.This study enrolled 3599 participants.No treatment was prescribed by this protocol and participants will be managed in accordance with normal medical practice.The planned total duration of the study was 10 years,with data being analyzed and reported every 2 years.Participants were assessed at nominal visits every 6 months and every effort was made to obtain as much of the required information as possible.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the final visit of the PROactive Study (NCT00174993).
* Willingness and ability to give written informed consent for the observational study.

Exclusion Criteria:

* There were no exclusion criteria.

Ages: 36 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk T2DM participants previously treated with pioglitazone and placebo in PROactive study (NCT00174993) were included in this study.
Sampling Method: Probability Sample
Enrollment: 3599 (Actual)
Dates: Start 2004-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- [Background] Erdmann E, Harding S, Lam H, Perez A. Ten-year observational follow-up of PROactive: a randomized cardiovascular outcomes trial evaluating pioglitazone in type 2 diabetes. Diabetes Obes Metab. 2016 Mar;18(3):266-73. doi: 10.1111/dom.12608. Epub 2016 Jan 8. PMID 26592506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 228 sites in 18 European countries including Austria, Belgium, Czech Republic, Denmark, Estonia, Finland, France, Germany, Hungary, Latvia, Lithuania, Netherlands, Norway, Poland, Slovakia, Sweden, Switzerland, and the United Kingdom from 02 November 2004 to 10 March 2015.
Pre-assignment Details: Participants with a historical diagnosis of Type 2 diabetes mellitus (T2DM) who were previously treated with pioglitazone or placebo in the PROactive study (NCT00174993) were enrolled in this observational study according to their originally assigned treatment group.
Groups:
- Pioglitazone: Participants who were previously treated with pioglitazone 15, 30, or 45 milligram tablets, orally, once daily during the PROactive study (NCT00174993) were followed up to 10 years in this observational study.
- Placebo: Participants who were previously treated with placebo-matching pioglitazone tablets, orally, once daily during the PROactive (NCT00174993) study were followed up to 10 years.
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 1820 | 1779
Completed | 932 | 907
Not Completed | 888 | 872
Not completed — Death | 619 | 649
Not completed — Withdrawal by Subject | 13 | 5
Not completed — Lost to Follow-up | 171 | 151
Not completed — Unconfirmed for lost to follow-up | 85 | 67

BASELINE CHARACTERISTICS:
Population: The observational study population consisted of participants who enrolled in this study after completing the final visit of PROactive study (NCT00174993).
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 1820 | 1779 | 3599
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (7.51) | 61.4 (7.80) | 61.6 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 632 | 626 | 1258
  Male | 1188 | 1153 | 2341
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1794 | 1760 | 3554
  Black | 7 | 3 | 10
  Asian/Oriental | 18 | 14 | 32
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: Participants]
  Austria | 45 | 47 | 92
  Belgium | 21 | 18 | 39
  Czech Republic | 40 | 40 | 80
  Denmark | 32 | 27 | 59
  Estonia | 50 | 53 | 103
  Finland | 138 | 124 | 262
  France | 28 | 30 | 58
  Germany | 104 | 104 | 208
  Hungary | 356 | 360 | 716
  Latvia | 178 | 175 | 353
  Lithuania | 120 | 115 | 235
  Netherlands | 16 | 18 | 34
  Norway | 44 | 47 | 91
  Poland | 374 | 366 | 740
  Slovakia | 39 | 42 | 81
  Sweden | 56 | 58 | 114
  Switzerland | 11 | 7 | 18
  United Kingdom | 168 | 148 | 316
Duration of T2DM [Mean (Standard Deviation); unit: Years] | 9.3 (6.81) | 9.3 (6.96) | 9.3 (6.88)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 87.72 (15.607) | 88.62 (15.451) | 88.17 (15.534)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 30.834 (4.7978) | 31.078 (4.7135) | 30.955 (4.7572)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With First Occurrence of Macro-vascular Event or Death
Description: The composite macro-vascular event or death included all-cause mortality, non-fatal myocardial infarction, cardiac intervention, stroke, major leg amputation (above the ankle), bypass surgery or revascularization in the leg. The percentage of participants in the observational study population having first occurrence of macro-vascular event or death during the 10-year observational study period was analyzed. The data were analyzed using the Cox regression with respect to time to the first occurrence of macro-vascular event or death.
Time Frame: Up to Year 10
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1820 | 1779
percentage of participants | 58 (NA) [NA to NA] | 60.3 (NA) [NA to NA]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test for statistical difference between pioglitazone and placebo with respect to time of first occurrence of the primary composite outcome event; Test type: Superiority or Other; p = 0.3444, Regression, Cox — No adjustment to the p-value; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.88 to 1.04]

2. Secondary Outcome: Incidences With Malignancies
Description: Percentage of participants with incidences of at least 1 malignancy was reported. All malignancies included adrenal, biliary, bladder, brain, breast, cervix, colon/rectal, gastric, hematological, hepatic, lung, mesothelioma, metastases, oesophageal, oropharyngeal, ovarian/uterine, pancreas, prostate, renal, skin and others.
Time Frame: Up to Year 10
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1820 | 1779
percentage of participants | 12.9 | 13.2
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.83 to 1.16]

ADVERSE EVENTS:
Description: Due to the observational nature of the study no safety data other than the monitored outcomes were collected.
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.